CLINICAL TRIAL: NCT00562289
Title: Closure of Patent Foramen Ovale or Anticoagulants Versus Antiplatelet Therapy to Prevent Stroke Recurrence
Brief Title: Patent Foramen Ovale Closure or Anticoagulants Versus Antiplatelet Therapy to Prevent Stroke Recurrence
Acronym: CLOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P060406
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-01

CONDITIONS: Ischemic Stroke; Patent Foramen Ovale; Atrial Septal Aneurysm; Migraine
Keywords: Stroke; Patent Foramen Ovale; Atrial septal aneurysm; Antiplatelet therapy; Oral anticoagulants; Transcatheter closure; Migraine
MeSH Terms: conditions — Ischemic Stroke; Foramen Ovale, Patent; Migraine Disorders; Stroke | interventions — Aspirin; Clopidogrel; Aspirin, Dipyridamole Drug Combination; antivitamins K; Rivaroxaban; Dabigatran; apixaban; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aspirin (Active Comparator): aspirin use like antiplatelet
  Interventions: Drug: aspirin
- anticoagulant (Experimental): Antivitamins K or rivaroxaban or dabigatran or apixaban
  Interventions: Drug: Antivitamins K or rivaroxaban or dabigatran or apixaban
- Devices for PFO closure (Experimental): Devices for PFO closure
  Interventions: Device: Devices for PFO closure

INTERVENTIONS:
Drug: aspirin — during the follow up
  Other Names: clopidogrel; combination aspirin-dipyridamole
  Arms: aspirin
Drug: Antivitamins K or rivaroxaban or dabigatran or apixaban — during the follow up
  Arms: anticoagulant
Device: Devices for PFO closure — endovascular treatment no longer than 21 days after the random.
  Other Names: Each device for PFO closure must have the CE mark; and be approved by the Interventional Cardiology Committee
  Arms: Devices for PFO closure

SUMMARY:
A patent foramen ovale (PFO) is found more frequently in patients with an ischemic stroke than in control subjects.

Therapeutic options to prevent stroke recurrence include antiplatelet drugs, oral anticoagulants, and transcatheter closure of the foramen. However, there are no published studies showing convincingly the superiority of any one of these strategies in preventing stroke recurrence.

The aim of this randomized clinical trial is to assess whether chronic anticoagulation on the one hand and transcatheter on the other hand are superior to chronic antiplatelet therapy in preventing stroke recurrence.

DETAILED DESCRIPTION:
Secondary prevention for stroke patients with PFO is a subject of considerable debate. Therapeutic options include antiplatelet drugs, oral anticoagulants, and transcatheter closure of the foramen. There are no published studies showing convincingly the superiority of any one of these strategies in preventing stroke recurrence. All the therapeutic options have some risks and unless randomised trials can define who should be treated with what (if anything), and for how long, we could end up exposing patients to unnecessary complications of treatment.

The primary objective of this study is to assess whether chronic anticoagulation (INR 2 to 3) on the one hand and endovascular treatment on the other hand are superior to chronic antiplatelet therapy in preventing stroke recurrence in young (16 to 60 years) patients with a PFO (> 30 microbubbles or associated with an atrial septal aneurysm) and an otherwise unexplained ischaemic stroke.

Secondary objectives of the study are:

* to evaluate the safety of the three therapeutic options, in terms of major drug-, device- or procedure-related complications, in order to allow a benefit/risk assessment of each therapeutic option in this population.
* to assess the rate of technical success and effectiveness of endovascular procedure to treat PFO and ASA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 16 <= age <= 60 ans.
* Recent (<= 6 months) ischemic stroke documented by CT-san or MRI (whatever the duration of symptoms: shorter or longer than 24 hours).
* Modified Rankin score <=3.
* Absence of any other identifiable cause of stroke
* Presence of a PFO with at least one of the following characteristics:

  * right-to-left shunt > 30 microbubbles, at rest or during provocative manoeuvres, by TTE ou TOE
  * associated ASA (base ≥ à 15 mm, total excursion > à 10 mm) by TOE
* Informed consent.

Exclusion Criteria:

* Any identifiable cause of ischemic stroke other than PFO.
* Isolated atrial septal defect or atrial septal defect associated with PFO with significant left-to-right shunt requiring closure.
* Previous surgical or endovascular treatments of PFO or ASA.
* Known or suspected pregnancy (beta hCG test must be performed before inclusion).
* Women who are breast-feeding.
* Inability to comply with the treatments or follow-up requirements of the study.
* No affiliation to the national health service.
* Presence of other medical problems that would either lead to inability to complete the trial or interfere with the assessment of outcomes.
* Participation in another study.
* Unable to understand the full meaning of the informed consent.
* Related medical treatments of the trial:

  * Long-term oral anticoagulation or antiplatelet therapy is indicated for another disease.
  * Contra-indication to antiplatelet therapy or oral anticoagulants :

    * 3-arm trial : contra-indication to aspirin or clopidogrel or antivitamins K
    * 2-arm trial (closure vs antiplatelet therapy) : contra-indication to aspirin or clopidogrel
    * 2-arm trial (antivitamins K vs antiplatelet therapy : contra-indication to antivitamins K or to any antiplatelet drug
  * Increased risk of bleeding, such as severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy, history of severe systemic bleeding (e.g. gastrointestinal bleeding, gross hematuria, intraocular bleeding, hemorrhagic stroke, or intracranial hemorrhage), or other history of bleeding diathesis or coagulopathy.
* Related to endovascular treatments :

  * Infection requiring antibiotics (inclusion is possible after healing, 4 weeks after withdrawal of antibiotics).
  * Very large or multi-perforated ASA for which endovascular treatments is deemed too risky.
  * Presence of thrombus or occlusion between the venous access and the right atrium.
  * Presence of an inferior vena cava filter.
  * Severe pulmonary hypertension.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 664 (Actual)
Dates: Start 2007-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
stroke(fatal or not) | during the follow up (between 2 or 9 years)

SECONDARY OUTCOMES:
Disabling stroke | during the follow-up
Ischemic stroke | during the follow-up
Cerebral haemorrhage | during the follow-up
Ischemic stroke, TIA, or systemic embolism | during the follow-up
Death (all causes) | during the follow-up
Vascular death | during the follow-up
Moderate to severe bleeding complications | during the follow-up
Procedural or device complications | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: MAS Jean-Louis, MD, PhD, Principal Investigator — Centre hospitalier sainte Anne
Locations (1):
- Hôpital Saint-Anne, Paris, France

REFERENCES:
- [Result] Mas JL, Derumeaux G, Guillon B, Massardier E, Hosseini H, Mechtouff L, Arquizan C, Bejot Y, Vuillier F, Detante O, Guidoux C, Canaple S, Vaduva C, Dequatre-Ponchelle N, Sibon I, Garnier P, Ferrier A, Timsit S, Robinet-Borgomano E, Sablot D, Lacour JC, Zuber M, Favrole P, Pinel JF, Apoil M, Reiner P, Lefebvre C, Guerin P, Piot C, Rossi R, Dubois-Rande JL, Eicher JC, Meneveau N, Lusson JR, Bertrand B, Schleich JM, Godart F, Thambo JB, Leborgne L, Michel P, Pierard L, Turc G, Barthelet M, Charles-Nelson A, Weimar C, Moulin T, Juliard JM, Chatellier G; CLOSE Investigators. Patent Foramen Ovale Closure or Anticoagulation vs. Antiplatelets after Stroke. N Engl J Med. 2017 Sep 14;377(11):1011-1021. doi: 10.1056/NEJMoa1705915. PMID 28902593
- [Derived] Turc G, Lee JY, Brochet E, Kim JS, Song JK, Mas JL; CLOSE and DEFENSE-PFO Trial Investigators. Atrial Septal Aneurysm, Shunt Size, and Recurrent Stroke Risk in Patients With Patent Foramen Ovale. J Am Coll Cardiol. 2020 May 12;75(18):2312-2320. doi: 10.1016/j.jacc.2020.02.068. PMID 32381162
- [Derived] Turc G, Calvet D, Guerin P, Sroussi M, Chatellier G, Mas JL; CLOSE Investigators. Closure, Anticoagulation, or Antiplatelet Therapy for Cryptogenic Stroke With Patent Foramen Ovale: Systematic Review of Randomized Trials, Sequential Meta-Analysis, and New Insights From the CLOSE Study. J Am Heart Assoc. 2018 Jun 17;7(12):e008356. doi: 10.1161/JAHA.117.008356. PMID 29910193
- [Derived] Mas JL, Derumeaux G, Amarenco P, Arquizan C, Aubry P, Barthelet M, Bertrand B, Brochet E, Cabanes L, Donal E, Dubois-Rande JL, Durand-Zaleski I, Ernande L, Finet G, Fraisse A, Giroud M, Guerin P, Habib G, Juliard JM, Leys D, Lievre M, Lusson JR, Marcon F, Michel P, Moulin T, Mounier-Vehier F, Pierard L, Piot C, Rey C, Rodier G, Roudaut R, Schleich JM, Teiger E, Turc G, Vuillier F, Weimar C, Woimant F, Chatellier G; CLOSE investigators. close: Closure of patent foramen ovale, oral anticoagulants or antiplatelet therapy to prevent stroke recurrence: Study design. Int J Stroke. 2016 Aug;11(6):724-32. doi: 10.1177/1747493016643551. Epub 2016 Apr 7. PMID 27056964